CLINICAL TRIAL: NCT02903784
Title: The Neural Basis of Language: A New Lighting. Study of Semantic Processing in MRI Mutimodale and Direct Electrical Stimulation
Brief Title: Neural Basis of Language Processing
Acronym: BNL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8674
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2011-05

CONDITIONS: Oligoastrocytoma; Astrocytoma; Oligodendroglioma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma | interventions — Magnetic Resonance Imaging; Diffusion Tensor Imaging; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- grade 2 glioma (Other): Patient with grade 2 glioma use a neuropsychological examination and brain imaging (fMRI and tractography)
  Interventions: Device: fMRI; Procedure: tractography; Other: neuropsychological examination
- healthy volunteers (Other): healthy volunteers use a neuropsychological examination and brain imaging (fMRI and tractography)
  Interventions: Device: fMRI; Procedure: tractography; Other: neuropsychological examination

INTERVENTIONS:
Device: fMRI — Patient with grade 2 glioma and healthy volunteers use a brain imaging (fMRI)
Procedure: tractography — Patient with grade 2 glioma and healthy volunteers use a brain imaging (tractography)
Other: neuropsychological examination — Patient with grade 2 glioma and healthy volunteers use a neuropsychological examination

SUMMARY:
According to the O.M.S. Classification, grade 2 glioma is a pre-cancerous lesion, slowly progressive, infiltrating the central nervous system, mainly affecting young adults.

This surgery should nevertheless be conducted in awake condition to achieve two conflicting goals: get maximum brain tissue infiltrated by the tumor while preserving the integrity of functional structures. So awake after opening the skull, the patient undergoes a series of preoperative tests, administered by a speech therapist present in the operating room. This procedure allows the neurosurgeon to establish an individual functional brain mapping in real time, through the observation by the SLP of the patient's answers to direct electrical stimulation applied to the cortical and sub-cortical. This support is based on the extraordinary plasticity demonstrated by the brain in the presence of a slowly progressive lesion. To ensure the patient the highest achievable load should increase our understanding of brain function, including the neural bases of language, glioma grade 2 is predominantly localized functional area of language.

DETAILED DESCRIPTION:
According to the O.M.S. Classification, grade 2 glioma is a pre-cancerous lesion, slowly progressive, infiltrating the central nervous system, mainly affecting young adults. Surgical excision of the tumor is the most appropriate care, with or without chemotherapy or radiotherapy.

This surgery should nevertheless be conducted in awake condition to achieve two conflicting goals: get maximum brain tissue infiltrated by the tumor while preserving the integrity of functional structures. So awake after opening the skull, the patient undergoes a series of preoperative tests (motor, sensory and / or language), administered by a speech therapist present in the operating room. This procedure allows the neurosurgeon to establish an individual functional brain mapping in real time, through the observation by the SLP of the patient's answers to direct electrical stimulation applied to the cortical and sub-cortical. This support is based on the extraordinary plasticity demonstrated by the brain in the presence of a slowly progressive lesion. To ensure the patient the highest achievable load should increase our understanding of brain function, including the neural bases of language, glioma grade 2 is predominantly localized functional area of language. Many studies apply to highlight the cortical organization of language, but the study of subcortical beams involved in this function, especially in the semantic language processing, has so far received less attention .

The use of electric direct intraoperative stimulation helps highlight the cortico-subcortical networks involved in language processing.

The new imaging techniques allow us to better understand the functional brain anatomy: the Diffusion Tensor can view the white matter bundles based on the diffusion of water molecules, functional MRI to visualize areas cortical functional.

ELIGIBILITY:
Inclusion Criteria:

Patients carry a grade glioma 2 functional area of language and presenting the information to receive surgical care provided in awake for the first time.

or Healthy volunteers will be selected using a matching age and sex of patients in the study (matched to a patient on two of the first forty patients).

Exclusion Criteria:

* Subject presenting cons-indications to MRI (ventricular shunt valve, ferromagnetic foreign bodies, pacemaker, implantable defibrillators, cochlear hearing implant, claustrophobia, ....)
* History of head trauma, ischemic stroke or intracerebral hematoma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
functional score | 1 day
  The intraoperative testing is performed by an evaluator (speech / neuropsychologist), present in the operating room, the patient's side. Its role is to identify functional disturbances induced by direct electrical stimulation.
  To do this, two standardized tests are administered to the patient alternately for the duration of the awake period. These tests are presented on a computer screen in PowerPoint format, with a picture every four seconds.

SECONDARY OUTCOMES:
Evaluation orthophonic | 1 day
  * Spontaneous Speech
  * Test oral denomination: DO. 80 with computerized measurement of reaction time
  * Verbal Fluence
    * Categorical: animals
    * Formal: letter / p /
  * Test semantic matching: PPTT with computerized measurement of the reaction time
  * trial test semantics / phonology
  * Image Designation
Evaluation orthophonic | 5 day
  * Spontaneous Speech
  * Test oral denomination: DO. 80 with computerized measurement of reaction time
  * Verbal Fluence
    * Categorical: animals
    * Formal: letter / p /
  * Test semantic matching: PPTT with computerized measurement of the reaction time
  * trial test semantics / phonology
  * Image Designation
Evaluation orthophonic | 3 month
  * Spontaneous Speech
  * Test oral denomination: DO. 80 with computerized measurement of reaction time
  * Verbal Fluence
    * Categorical: animals
    * Formal: letter / p /
  * Test semantic matching: PPTT with computerized measurement of the reaction time
  * trial test semantics / phonology
  * Image Designation
Imagery Data | 1 day
  Imagery Data
Imagery Data | 5 day
  Imagery Data
Imagery Data | 6 month
  Imagery Data

IPD SHARING:
Plan to Share IPD: Undecided